CLINICAL TRIAL: NCT07335484
Title: Prospective, Multicenter, Single Arm Feasibility and Safety Study of the Axonics External Trial System (ETS-02)
Brief Title: Aquarius Pilot Study to Evaluate the New Axonics Trial System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Axonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-0179
Record Dates: First submitted 2026-01-06; First posted 2026-01-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Urinary Urge Incontinence (UUI); Urinary Frequency (UF); Fecal Incontinence (FI); Overactive Bladder (OAB)
Keywords: Peripheral nerve evaluation; External trial system; Pilot study
MeSH Terms: conditions — Urinary Incontinence, Urge; Fecal Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Patients diagnosed with OAB and/or FI who are candidates for Axonics SNM (PNE) procedure (Experimental): External trial system used evaluated whether patients with OAB or FI will be responsive to sacral neuromodulation.
  Interventions: Device: Axonics External Trial System (ETS)

INTERVENTIONS:
Device: Axonics External Trial System (ETS) — A temporary electrode wire is passed through the S3 foramen with or without fluoroscopic guidance. The wire is then connected to an external pulse generator (EPG) and is worn for a trial period ranging from 3-7 days.
  Other Names: Basic or Advanced Trial

SUMMARY:
Evaluation of the new Axonics External Trial System (ETS-02) in patients with overactive bladder (OAB) and/or fecal incontinence (FI).

DETAILED DESCRIPTION:
The trial system is used to determine if patients are responsive to sacral neuromodulation (SNM) prior to receiving the Axonics implantable neurostimulator (INS) which is approved for the treatment of OAB and FI. This study is evaluating the feasibility and safety of the new Axonics External Trial System (ETS-02) in patients with overactive bladder (OAB) and/or fecal incontinence (FI).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Provides written informed consent prior to trial procedures
* Primary indication of OAB (UUI/UF) or chronic FI who are considered candidates for an Axonics PNE procedure as assessed by the physician per product IFU

Exclusion Criteria:

* Any participant that the study Investigator deems to be a poor candidate for any reason, including, but not limited to, inability to complete a baseline bladder or bowel diary or to be compliant with study visits
* Planned changes to current regimen of medications during the trial period that could impact bladder or bowel function
* Current urinary tract mechanical obstruction (e.g., benign prostatic enlargement or urethral stricture)
* Current symptomatic urinary tract infection (UTI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Feasibility | Day 5-7
  Trial system success rate, defined as the proportion of participants with the Axonics ETS still attached and operable end of the trial period.
Adverse Events reporting (Safety) | Day 0-7
  Device- or procedure-related adverse events as determined by the independent physician adjudicated (IPA).

CONTACTS AND LOCATIONS:
Overall Officials: Ailsa Wilson Edwards, MD, Principal Investigator — Calvary North Adelaide Hospital

IPD SHARING:
Plan to Share IPD: No